CLINICAL TRIAL: NCT01365884
Title: Proof of Concept Study for First-Sight Refractive Error Correction: Direct Comparison to Autorefraction Results in Children 7 to 18 Years of Age
Brief Title: First-Sight Refractive Error Correction: Direct Comparison to Autorefraction Results in Children 7 to 18 Years of Age
Status: Terminated | Type: Observational
Why Stopped: Low subject recruitment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0201-11-FB
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Proof of concept study to compare the best corrected visual acuity obtained via First-Sight lenses with the autorefraction in children.

DETAILED DESCRIPTION:
Uncorrected refractive error is a frequent cause of visual impairment in children most prevalent in rural or underserved areas in the global population. In 2006, the World Health Organization released global estimates on visual impairment. According to their findings, there are approximately 314 million people in the world whose vision is impaired. Of this population 90% of those individuals live in developing countries and 153 million cases are believed to be due to uncorrected refractive error. Children, ages five to 15 years, suffer from refractive errors (mostly myopia, hyperopia, and astigmatism) that can be improved to normal vision. It is estimated that by 2020, approximately one third of the world's population (2.5 billion) will be affected by myopia alone14. The prevalence of refractive error in school-aged children is significant especially the impact on a child's life in terms of education and development.

Studies in Western populations have collectively shown that myopia occurs <5% in children 8 years and younger. Sampling studies in other countries worldwide have shown that there is higher prevalence of myopia among Southeast Asia children and less among Australian children.1-11 Refractive error study in Eastern Nepal found 2.9% of children had vision of 20/40 or worse of which 56% of the 200 eyes tested was caused by refractive error due to myopia, hyperopia and astigmatism.12

The challenge is to determine the most effective and accessible method of detecting refractive error and dispensing spectacles for better vision. Children who have access to clinical setting typically receive prescriptive spectacles to correct refractive errors. However, in underserved areas where standard eye care may be absent, children are unable to receive the benefits of normal or near normal vision. The challenge is to determine the most effective and accessible method of detecting refractive error and dispensing spectacles for better vision

In the clinical setting, refractive error is corrected by prescribing spectacles or contact lenses on a daily basis. Typically the patient will first undergo autorefraction, in which a computer-controlled machine objectively calculates the refractive error present as a starting point for the subjective refraction test. This machine, however, is cumbersome and not easily transportable abroad. Typically the machine is held up to the patient's forehead and they are asked to look into the machine at a distant object. While they are looking at this object the machine calculates the refractive error.

First-Sight is a simplified way to correct refractive error. It is easily portable, making it accessible to remote areas of the world. Unlike the study cited above, First-Sight can be taken to remote areas where clinics are not available and patients are not able to afford to pay for the clinic visit. As it is a simplified technique, local health care workers may easily be able to learn how to use First-Sight and dispense spectacles to those in need. Lastly, sponsors of First-Sight will provide the refracting kit and dispense custom-made spectacles at no cost to health care workers and children respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are between 7 to 18 years of age.
2. Healthy subjects
3. A refractive error of -4.50 to +4.50 diopter spherical error and astigmatism up to -1.50 diopters on manifest refraction and autorefraction as documented in their medical records.
4. Best corrected visual acuity (BCVA) of 20/20 with cycloplegic refraction.
5. No known ocular pathology from previous clinical exams that may limit best corrected visual acuity.

Exclusion Criteria:

1. Refractive error greater than -4.50 or +4.50 diopter, or astigmatism greater than -1.50 diopters.
2. Known ocular (corneal, lenticular, vitreal, or retinal) pathology that may limit BCVA.
3. Best corrected visual acuity with spectacles of 20/25 or worse.
4. Any previous surgical or laser procedures that may limit BCVA
5. Narrow angles of the eyes
6. Adults, 19 years or older

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population with refractive error between -4.50 to +4.50 diopter spherical error and astigmatism up to -1.50 diopters.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-08-05 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2014-02-12 (Actual)

PRIMARY OUTCOMES:
Compare refracting methods | 1 hour
  Will measure children's vision with First-Sight refracting kit and compare it to the two standard methods used in clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Feilmeier, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Ophthalmology, Omaha, Nebraska, United States